CLINICAL TRIAL: NCT00972361
Title: Routine Preoperative Hemostatic Laboratory Evaluation Prior to Tonsillectomy or Adenoidectomy in Children - a Necessity or Habitude?
Brief Title: Routine Preoperative Hemostatic Laboratory Evaluation Prior to Tonsillectomy or Adenoidectomy in Children
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 0134-08-EMC
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Coagulation Abnormalities
Keywords: Adenoidectomy; Tonsillectomy; Ventilation Tubes; Preoperational screening; Coagulation Profile; Lupus anticoagulant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Routine analysis of coagulation profile is recommended before adenoidectomy, tonsillectomy or ventilation tubes insertion in children.

A proportion of those children reveal borderline abnormal values of Partial Prothrombin Time (aPTT) or Prothrombin Time (PT) and then they are referred to a consultant hematologist for further evaluation and recommendations before surgery.

The purpose of this study is to summarize the causes of referrals in a cohort of 200 children and to assess the further laboratory analysis preformed and the results obtained.

DETAILED DESCRIPTION:
Data from about 200 children that were evaluated for abnormal coagulation tests performed before minor surgery.

The data will include cause of referral, laboratory analysis performed and results.

If the data allows the outcome of the operation and bleeding complications, will also recorded.

ELIGIBILITY:
Inclusion Criteria:

* All the patients referred to the pediatric hematology unit for evaluation due to coagulation abnormalities before minor surgery

Exclusion Criteria:

* No exclusion are applicable

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Data from about 200 children that were evaluated for abnormal coagulation tests performed before minor surgery.
  The data will include cause of referral, laboratory analysis performed and results.
  If the data allows the outcome of the operation and bleeding complications, will also recorded.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Principal Investigator — Pediatric Dpt B and Pediatric Hemaology Unit - Ha'Emek Medical Center - Afula - Israel
Locations (1):
- Pediatric Hematology Unit and Pediatric Dpt B - HaEmek Medical Center, Afula, Israel